CLINICAL TRIAL: NCT00467220
Title: Effect of Daily Calorie Restriction or Alternate-day Reductions in Calorie Intake on Risk for Cardiovascular Disease and Cancer
Brief Title: Effect of Daily Calorie or Alternate-day Calorie Reductions on Risk for Cardiovascular Disease and Cancer
Acronym: 1072
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H3049-30095-01; NIH-PPG (Other Grant/Funding Number: National Institutes of Health)
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Moderately Overweight Individuals
Keywords: Calorie restriction; alternate day fasting; calorie intake
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Subjects will follow all study tasks but will not be required to follow a calorie-restricted meal plan.
- Alternate Day Fasting Arm (Other): Subjects in this arm will be asked to alternate between one day of eating as they wish versus one day on a calorie-restricted meal plan. Subjects will follow this alternating meal plan for 3 months.
  Interventions: Behavioral: calorie restriction
- Calorie Restriction (Other): Subjects in this arm will be asked to follow a calorie-restricted meal plan, daily, for three months.
  Interventions: Behavioral: calorie restriction

INTERVENTIONS:
Behavioral: calorie restriction — Subjects in the "calorie restriction" arm and the "alternate day fasting" arm will be asked to follow a menu plan, for three months, that includes some level of calorie restriction.
  Arms: Alternate Day Fasting Arm; Calorie Restriction

SUMMARY:
The purpose of this study is to examine and compare the effects of alternate-day reductions in calorie intake or daily calorie restriction on the risk for cardiovascular disease and cancer.

DETAILED DESCRIPTION:
Overweight individuals are at greater risk for certain chronic diseases such as cardiovascular disease and cancer when compared to those who are normal weight. Dietary restriction has been shown to lower the risk of these chronic diseases in overweight human subjects as well as in normal weight rodents. The majority of studies examining dietary restriction protocols in rodents or humans implement daily calorie restriction (CR), i.e. where the amount of energy consumed is decreased by a certain percentage every day. Another dietary restriction regimen employed, although less commonly, is intermittent caloric restriction, or alternate-day fasting (ADF), i.e. where food is available ad-librium every other day, alternating with a partial or complete caloric restriction day. Recent findings suggest that ADF may modulate certain indices of disease risk to a similar extent as daily CR in animal models. The effect of ADF regimens in comparison with CR regimens on disease risk has yet to be performed in human subjects, however. ADF protocols need not result in weight loss, and would therefore be appropriate for non-obese individuals. Accumulating evidence suggest that adipose tissue may play a role in modulating chronic disease risk by releasing substrates, such as fatty acids, or a variety of hormones, including adiponectin and leptin. The effect of ADF and CR on adipose tissue metabolism and hormone release remains unclear. Accordingly, the aim of the present study is to compare ADF regimes to CR for their effects on risk factors for cardiovascular disease and cancer and their effects on adipose tissue metabolism and hormone secretion, in normal weight to modestly overweight (BMI 22-27 kg/m2) human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female; body mass index (BMI) between 20-30 kg/m2;
* Age between 35-65 years; sedentary (light exercise less than 1h per week) or moderately active (1 to 2h per week);
* Weight stable for >3 months prior to the beginning of the study;
* Able to give written informed consent;
* Female subjects must be post-menopausal for at least 2 years and can not be on hormone replacement therapy (HRT).

Exclusion Criteria:

* Diabetic;
* History of cardiovascular disease, i.e. myocardial infarction or stroke;
* History of cancer;
* Taking glucose lowering medication;
* Taking weight loss medication

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2015-12-17 (Actual); Study Completion 2015-12-17 (Actual)

PRIMARY OUTCOMES:
Adipose tissue dynamics | 12 weeks
  Parameters measured will include adipose tissue dynamics (triglyceride turnover, lipolysis, de novo lipogenesis, adipose cell proliferation), adipose tissue morphology (cell size and number), adipose tissue hormone levels (adiponectin, leptin), skin turnover (keratin dynamics), T-lymphocyte proliferation, as well as plasma lipid and lipoprotein, homocysteine, and C-reactive protein levels.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Hellerstein, MD, PhD, Principal Investigator — University of California, Berkeley; University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717